CLINICAL TRIAL: NCT00227422
Title: A Phase IV, Partially Double-blind Study to Demonstrate Non-inferiority of GSK Biologicals' Mencevax™ ACWY (New Process) Versus Mencevax™ ACWY (Current Process) When Administered as a Single Dose to Subjects Aged 2-30 Yrs
Brief Title: Assess the Non-inferiority of GSK Biologicals' Mencevax™ ACWY (Manufactured by a New Process) vs Mencevax™ ACWY (the Already Existing Vaccine in the Market) When Given as a Single Dose to Subjects Aged 2-30 Yrs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102394
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
Keywords: Neisseria meningitidis serogroups A & C diseases; Hib diseases
MeSH Terms: conditions — Meningococcal Infections | interventions — PsACWY vaccine

INTERVENTIONS:
Biological: Mencevax ACWY

SUMMARY:
The purpose of this study is to evaluate that the vaccine produced with the new process and administered as a single dose is at least as good as the existing Mencevax™ ACWY vaccine in terms of immunogenicity, safety and reactogenicity, in healthy subjects aged 2-30 years.

DETAILED DESCRIPTION:
"Randomized study with four groups to receive one of the following vaccination regimens: - One of the 3 lots of GSK Biologicals' Mencevax™ ACWY vaccine manufactured by the new process (3 different groups) - GSK Biologicals' already existing Mencevax™ ACWY

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female between 2 and 30 years of age at the time of vaccination.
* If the subject is female, she must be of non-childbearing potential. If a subject is a female of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after vaccination.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Vaccination with a meningococcal vaccine within the last five years.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 15 days before vaccine administration and ending 30 days after.
* History of or known exposure to meningococcal serogroup A, C, W135 or Y disease or contacts with subjects who had meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 324
Dates: Start 2005-06; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
1 month after vaccination, measurement of serum bactericidal titers against meningococcal serogroups A, C, W135 and Y (SBA-MenA; SBA-MenC; SBA-MenW135 and SBA-MenY)

SECONDARY OUTCOMES:
Immuno : the same immuno evaluation performed 1 month after vaccination will also be performed before vaccination; also vaccine response at Post-dose 1.
Safety : Solicited symptoms during day 0-3, unsol. symptoms during day 0-30 & SAEs during entire study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 102394 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102394 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102394 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102394 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102394 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102394 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register